CLINICAL TRIAL: NCT02454868
Title: Remifentanil Minimum Effective Dose for Children Intubation Without Neuromuscular Blockade
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brasilia University Hospital (Other)
Collaborators: University of Brasilia (Other)
Responsible Party: Principal Investigator, Gabriel Magalhaes Nunes Guimaraes, MSc, Brasilia University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UBrasilia
Record Dates: First submitted 2015-05-14; First posted 2015-05-27 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Underdosing of Unspecified General Anesthetics
Keywords: Remifentanil; Intubation; Children
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study arm (Experimental): There is a single study arm. Remifentanil will be infused before intubation. The first patient will receive remifentanil 2mg/kg. If a success occurs the next patient's dose will be decreased by 0.25mg/kg and else it will be increased by 0.25mg/kg. This rule will apply recursively as Dixon's Up-And-Down Method.
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — Remifentanil for intubation without neuromuscular blockade
  Other Names: Ultiva

SUMMARY:
Introduction: remifentanil's optimal dose for children intubation without neuromuscular blockade is unknown. Method: phase IV adaptative trial using Dixon's up-and-down method for modeling remifentanil's dose-response curve for adequate intubation conditions as defined by previous studies.

DETAILED DESCRIPTION:
Introduction: remifentanil's optimal dose for children intubation without neuromuscular blockade is unknown.

Method: phase IV adaptative trial using Dixon's up-and-down method for modeling remifentanil's dose-response curve for adequate intubation conditions as defined by previous studies. Remifentanil doses starting from 2mg/kg will be infused before intubation. When a success occurs next patient's dose will be decreased by 0.25mg/kg/h. When a success does not occur the next patient's dose will be increased by 0.25mg/kg/h. Intubation will be considered adequate if patient does not cough, does not move, if vocal cords are open, if larigocsocpic Cormack grade I or II.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II
* Scheduled for surgery under general anesthesia.

Exclusion Criteria:

* Predicted difficult airway
* Severe neurologic or cardiologic conditions
* Recent upper airway infectious diseases

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2016-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Adequate intubation condition (dichotomic) as an assessment of success rate | intraoperative
  Intubation is adequate if patient does not cough, does not try to breathe, vocal cords do not move, patient does not react and laringoscopy is Cormack class I or II

CONTACTS AND LOCATIONS:
Overall Officials: Catia S Goveia, MSc, Principal Investigator — University of Brasilia

REFERENCES:
- [Derived] Ono AH, Moura TR, Goveia CS, Guimaraes GMN, de Araujo Ladeira LC, da Silva HBG. ED50 of remifentanil for providing excellent intubating conditions when co-administered with a single standard dose of propofol without the use of muscle relaxants in children: dose-finding clinical trial. J Anesth. 2018 Aug;32(4):493-498. doi: 10.1007/s00540-018-2502-z. Epub 2018 May 4. PMID 29728755